CLINICAL TRIAL: NCT00235703
Title: Inter-Mountain Project on Antimicrobial Resistance and Therapy (IMPART)
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Other Study IDs: RS1/CCR820631-01
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2005-10

CONDITIONS: Upper Respiratory Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Device: Antimicrobial Prescribing Decision Support

SUMMARY:
This is a four-year study, funded by the Center for Disease Control and Prevention, related to antimicrobial resistance in rural communities. The project consists of four components: A) surveillance of antimicrobial resistance, B) promotion of appropriate antimicrobial drug prescribing, C) preliminary assessment of the environmental impact of antimicrobials, and D) the development of new antimicrobial products. Six rural communities in Utah, and six rural communities in Idaho are participating in this study. Component D is being performed by investigators at Harvard University, under the direction of Co-Investigator Roger Inouye.

ELIGIBILITY:
Inclusion Criteria:

* Suspected upper respiratory infection patients in 12 rural communities in Utah and Idaho

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13000
Dates: Start 2001-10; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Samore, MD, Principal Investigator — University of Utah

REFERENCES:
- [Result] Samore MH, Bateman K, Alder SC, Hannah E, Donnelly S, Stoddard GJ, Haddadin B, Rubin MA, Williamson J, Stults B, Rupper R, Stevenson K. Clinical decision support and appropriateness of antimicrobial prescribing: a randomized trial. JAMA. 2005 Nov 9;294(18):2305-14. doi: 10.1001/jama.294.18.2305. PMID 16278358